CLINICAL TRIAL: NCT03400475
Title: The Use of Topical Subgingival Application of Simvastatin Gel in the Treatment of Peri-Implant Mucositis: A Pilot Study
Brief Title: Use of Topical Subgingival Application of Simvastatin Gel in the Treatment of Peri-Implant Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ahmed Mohamed Mahrous (Other)
Collaborators: Greater New York Academy of Prosthodontics (Unknown); American College of Prosthodontists Education Foundation (Unknown); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Mahrous, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201410714
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Results first posted 2018-11-29 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Peri-implant Mucositis
Keywords: topical; subgingival; simvastatin
MeSH Terms: interventions — Simvastatin; Lecithins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the study coordinator will know whether the intervention is simvastatin or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin group (Treatment) (Experimental): Will receive 0.1 ml prepared Simvastatin in 1.2% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri-implant gingival sulcus using a plastic syringe with a blunt cannula.
  Interventions: Drug: Simvastatin
- Control group (Placebo Comparator): Will receive a placebo of 0.1 ml 40% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri-implant gingival sulcus using a plastic syringe with a blunt cannula.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Simvastatin — One topical application in peri-implant gingival crevice
  Other Names: Simvastatin Powder U.S.P.
  Arms: Simvastatin group (Treatment)
Other: Placebo — One topical application in peri-implant gingival crevice
  Other Names: Lecithin/isopropyl palmitate solution, Poloxamer 407 gel; Lipoil®, Polox Gel 20%®
  Arms: Control group

SUMMARY:
This study seeks to test the recently discovered anti-inflammatory action of statins on inflamed mucosa surrounding dental implants.

Hypothesis: The application of 1.2% simvastatin gel will decrease peri-implant inflammation.

The pilot study will involve 44 subjects divided into a test and control group. The test group shall receive topical simvastatin gel administered around the implant with a blunt tipped needle. The control group will receive a placebo.

Inflammatory state shall be determined at baseline as well as follow up visits at 24 hours, 1 week, and 1 month by clinical indices of inflammation as well as biochemical markers of inflammation gathered from around the implants.

DETAILED DESCRIPTION:
Following signing the consent document the following will occur:

1. Screening Patients will complete standard medical and dental health history forms, followed by a study specific screening questionnaire. if the patient is deemed eligible, the patient will be examined clinically. The clinical examination will include diagnostic procedures typical of an implant recall visit. Initially, the sulcus will be probed with a periodontal probe; if bleeding on probing is elicited, then a radiograph will be made.

   The following shall be done to screen the patients:
   1. Periapical radiographs of the implant to determine bone loss, if bone loss is found the patient will be excluded from the study.
   2. Bleeding on probing will be assessed by using a periodontal probe passed along the gingival crevice, and bleeding scores will be assessed passing the probe with a force of 0.25 N.
   3. If a woman is of childbearing age and suspected of being pregnant, a urine pregnancy test shall be made at this time.

   If the patient exhibits no bleeding on probing, or signs of mesial/distal bone loss greater than 1mm from the accepted reference point on the implant system the patient will be excluded from the study.
2. Subject allocation

   Subjects will be assigned with equal allocation into the following groups:
   1. Test group: will receive 0.1 ml prepared Simvastatin in 1.2% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri-implant gingival sulcus using a plastic syringe with a blunt cannula.
   2. Control group: will receive a placebo of 0.1 ml 40% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri implant gingival sulcus using a plastic syringe with a blunt cannula.
3. Baseline measurements Baseline measurements will be made at least 48 hours after screening (allowing time for complete hemostasis of peri-implant crevicular mucosa after bleeding induced by probing in the screening visit).

   Following baseline measurements, Test and Control interventions will be administered.

   The baseline measurements include the following:
   1. Peri-implant crevicular fluid (PICF) collection: Each implant site will be isolated with cotton rolls and light air will be applied over the side to eliminate ambient salivary contamination of the PICF sample. Sampling will be done using paper strips that are inserted with cotton forceps into the gingival crevice until mild resistance is felt. After gingival crevicular fluid (GCF) collection, the volumes are immediately quantified using the Periotron 8000 instrument.
   2. Gingival Index: Using the Gingival index by Loe and Sillness 1963, the inflammatory state of the buccal, lingual, mesial and distal surfaces of the gingiva will be scored using the following score system:

      0= normal gingival without signs of inflammation, no inflammation, no bleeding
      1. minor inflammation , slight discoloration, minor surface alterations, no bleeding
      2. moderate inflammation, redness, swelling, bleeding upon probing and under pressure
      3. strong inflammation, strong redness and swelling, tendency toward spontaneous bleeding, ulcerations After a score is given to each site, the scores will be summed together and divided by 4 to reach an overall score.
   3. Probing depth: Measured by a calibrated periodontal probe at 6 different locations, mesiobuccal, midbuccal, distobuccal, distolingual, midlingual, and mesiolingual.
4. Administration of test and control intervention will be delivered into the peri- implant gingival sulcus using a plastic syringe with a blunt cannula following baseline measurements. 0.1ml of gel will be administered with a blunt cannula evenly distributed in the peri-implant sulcus. The investigator will not know whether the subject is receiving the active or control intervention.
5. Recall appointments and measurements Both Test and Control subjects will be scheduled recall visits. Recalls will be done at 24 hours (+ or - 3 hours), 1 week (+ or - 12 hours), and 1 month (+ or - 11 days).

   On each recall visit, the following procedures will take place:
   1. PICF collection: procedures identical to those performed on the baseline visit
   2. Gingival index recording: Identical to that performed on the baseline visit
   3. probing depth measurement : procedures identical to that performed at the baseline visit * these measurements will be made by a blinded investigator
6. Cytokine analysis Due to study constraints, not all PICF samples collected from subjects will be analyzed in the pilot study. The samples that will be analyzed will be selected randomly from the study population. Cytokine samples from only 13 randomly selected subjects from the test group, as well as 13 randomly selected subjects from the control group will be analyzed. Of these randomly selected samples, only those collected at baseline, 24 hours, and at 1 week will be analyzed. The remaining cytokine samples will be evaluated as part of a later study. Cytokine quantities will be determined using; a commercial 22 multipixed fluorescent bead based immunoassay and luminex 100 IS instrument. The kit used is the MILLIPLEX map Human Cytokine/ Chemokine Magnetic Bead Panel- Immunology Multiplex Assay (HCYTOMAG-60K) capable of detecting IL-1Beta;, TNF-Alpha;, IL-6, IL-8.

The study in total will take 1 month and 2 days. All visits will generally take 0.5-1.5 hours. No long term follow up will be required.

ELIGIBILITY:
Inclusion Criteria:

* Read, understand, and sign the informed consent forms
* Have at least 1 dental implant
* Have no evidence of peri-implantitis as evidenced by mesial and distal bone loss more than 1 mm from the accepted reference point round the implants on the periapical radiograph
* Demonstrate peri-implant mucositis as evidenced by bleeding on probing with 0.25 N/cm

Exclusion Criteria:

* Have allergic reactions to simvastatin
* Have peri-implantitis as evidenced by more than 1 mm of mesial and distal bone loss from an accepted reference point on the implants on the periapical radiograph
* Demonstrate no bleeding on probing with 0.25 N/ cm
* Have uncontrolled systemic disease
* Pregnancy or females who suspect/may be pregnant, as well as nursing and breast feeding mothers
* Take statin / HMG-CoA reductase inhibitor medications
* Smokers
* Require antibiotic prophylaxis
* Take anti-inflammatory medication, immunosuppressive medications or immunosuppressed patients
* Have paraben allergies
* Have soybean allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mahrous, B.D.S., M.S., Principal Investigator — University of Iowa College of Dentistry and Dental Clinics
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradeep AR, Thorat MS. Clinical effect of subgingivally delivered simvastatin in the treatment of patients with chronic periodontitis: a randomized clinical trial. J Periodontol. 2010 Feb;81(2):214-22. doi: 10.1902/jop.2009.090429. PMID 20151799
- [Background] Liskmann S, Vihalemm T, Salum O, Zilmer K, Fischer K, Zilmer M. Correlations between clinical parameters and interleukin-6 and interleukin-10 levels in saliva from totally edentulous patients with peri-implant disease. Int J Oral Maxillofac Implants. 2006 Jul-Aug;21(4):543-50. PMID 16955604
- [Background] Konttinen YT, Lappalainen R, Laine P, Kitti U, Santavirta S, Teronen O. Immunohistochemical evaluation of inflammatory mediators in failing implants. Int J Periodontics Restorative Dent. 2006 Apr;26(2):135-41. PMID 16642902
- [Background] Sakoda K, Yamamoto M, Negishi Y, Liao JK, Node K, Izumi Y. Simvastatin decreases IL-6 and IL-8 production in epithelial cells. J Dent Res. 2006 Jun;85(6):520-3. doi: 10.1177/154405910608500608. PMID 16723648
- [Background] Guncu GN, Akman AC, Gunday S, Yamalik N, Berker E. Effect of inflammation on cytokine levels and bone remodelling markers in peri-implant sulcus fluid: a preliminary report. Cytokine. 2012 Aug;59(2):313-6. doi: 10.1016/j.cyto.2012.04.024. Epub 2012 May 14. PMID 22592038
- [Background] Duarte PM, de Mendonca AC, Maximo MB, Santos VR, Bastos MF, Nociti Junior FH. Differential cytokine expressions affect the severity of peri-implant disease. Clin Oral Implants Res. 2009 May;20(5):514-20. doi: 10.1111/j.1600-0501.2008.01680.x. Epub 2009 Mar 11. PMID 19302394
- [Background] Ferro D, Parrotto S, Basili S, Alessandri C, Violi F. Simvastatin inhibits the monocyte expression of proinflammatory cytokines in patients with hypercholesterolemia. J Am Coll Cardiol. 2000 Aug;36(2):427-31. doi: 10.1016/s0735-1097(00)00771-3. PMID 10933353

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: Will receive 0.1 ml prepared Simvastatin in 1.2% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri-implant gingival sulcus using a plastic syringe with a blunt cannula.
  Simvastatin: One topical application in peri-implant gingival crevice
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 24 | 22
Completed | 24 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: each patient is considered one unit
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.45 (13.3) | 63.1 (14.3) | 63.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin 1 B at Base to 24 Hours
Description: Measuring the change in Cytokine levels in the peri implant crevicular fluid ( Fluid around the implant) by extracting the fluid and measuring the levels of the interlukins in the fluids in Micrograms per dicileter ( ug/dl)
Time Frame: Baseline- 24hrs
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Groups:
- Simvastatin Group ( Treatment ): Will receive 0.1 ml prepared Simvastatin in 1.2% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri-implant gingival sulcus using a plastic syringe with a blunt cannula.
  Simvastatin: One topical application in peri-implant gingival crevice
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | -1.075 (15.587) | 1.013 (5.273)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2.088

2. Primary Outcome: Change in Interleukin 1 B at Base to 1 Week
Description: as for outcome 1
Time Frame: Baseline - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 2.5016 (15.4701) | -1.095 (8.6050)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.59

3. Primary Outcome: Change in Interleukin 1 B 24 Hours - 1 Week
Description: as for outcome 1
Time Frame: 24 hours - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 3.577 (14.137) | -2.108 (10.569)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.596

4. Primary Outcome: Change in Interleukin 6 at Base to 24 Hours
Description: as for outcome 1
Time Frame: Baseline - 24 hours
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 0.118 (0.954) | 0.201 (0.880)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.083

5. Primary Outcome: Change in Interleukin 6 Baseline to 1 Week
Description: as for outcome 1
Time Frame: Baseline - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 0.304 (1.3744) | 0.275 (1.296)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.581

6. Primary Outcome: Change in Interleukin 6 24 Hours - 1 Week
Description: as for outcome 1
Time Frame: 24 hours - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 0.185 (2.039) | 0.073 (1.522)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.029

7. Primary Outcome: Change in Interleukin 8 at Base to 24 Hours
Description: as for outcome 1
Time Frame: Baseline - 24 hours
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 0.00 (331.021) | 64.696 (197.902)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -64.696

8. Primary Outcome: Change in Interleukin 8 at Base to 1 Week
Description: as for outcome 1
Time Frame: Baseline - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 131.368 (480.835) | 20.275 (389.666)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 111.03

9. Primary Outcome: Change in Interleukin 8 24 Hours to 1 Week
Description: as for outcome 1
Time Frame: 24 hours - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 168.894 (548.154) | -44.42 (484.019)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 213.314

10. Primary Outcome: Change in Tumor Necrosis Factor Alpha at Base to 24 Hours
Description: as for outcome 1
Time Frame: Baseline- 24hrs
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 37.526 (1.266) | -0.17 (1.589)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 37.356

11. Primary Outcome: Change in Tumor Necrosis Factor Alpha at Base to 1 Week
Description: as for outcome 1
Time Frame: Baseline - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 1.5833 (5.665) | -0.0704 (2.8536401)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.6537

12. Primary Outcome: Change in Tumor Necrosis Factor Alpha 24 Hours to 1 Week
Description: as for outcome 1
Time Frame: 24hrs - 1 week
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (ug/dl)
Arm/Group | Simvastatin Group ( Treatment ) | Control Group
Number analyzed (Participants) | 24 | 22
Micrograms per deciliter (ug/dl) | 1.641 (5.7217) | 0.095 (3.633)
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment ) vs Control Group; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.552

13. Secondary Outcome: Gingival Index Level (Derived From an Average Over the 4 Implant Sites) at Baseline
Description: Using the Gingival index by Loe and Sillness 1963, the inflammatory state of the Buccal, Lingual, Mesial and Distal Surfaces of the gingiva will be scored using the following score system:
  0= normal gingival without signs of inflammation, no inflammation, no bleeding
  1. minor inflammation , slight discoloration, minor surface alterations, no bleeding
  2. moderate inflammation, redness, swelling, bleeding upon probing and under pressure
  3. strong inflammation, strong redness and swelling, tendency toward spontaneous bleeding, ulcerations After a score is given to each site the scores are summed together and divided by 4 to reach an overall score.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Simvastatin Group ( Treatment): Will receive 0.1 ml prepared Simvastatin in 1.2% (W/V) Lecithin/isopropyl palmitate solution (Lipoil®), Poloxamer 407 gel (Polox Gel 20%®) applied topically into the peri-implant gingival sulcus using a plastic syringe with a blunt cannula.
  Simvastatin: One topical application in peri-implant gingival crevice
Arm/Group | Simvastatin Group ( Treatment) | Control Group
Number analyzed (Participants) | 24 | 22
participants
  Gingival index score of 0.50 | 1 | 0
  Gingival index score of 1 | 0 | 0
  Gingival index score of 1.25 | 18 | 12
  Gingival index score of 1.5 | 4 | 8
  Gingival index score of 1.75 | 1 | 2
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment) vs Control Group; Test type: Superiority; p = 0.071, Fisher Exact

14. Secondary Outcome: Gingival Index Level (Derived From an Average Over the 4 Implant Sites) at 24 Hours
Description: as for outcome 13
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Simvastatin Group ( Treatment) | Control Group
Number analyzed (Participants) | 24 | 22
participants
  Gingival sscore of 0.50 | 1 | 1
  Gingival sscore of 1 | 16 | 4
  Gingival sscore of 1.25 | 6 | 12
  Gingival sscore of 1.50 | 1 | 5
  Gingival sscore of 1.75 | 0 | 0
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment) vs Control Group; Test type: Superiority; p = 0.071, Fisher Exact

15. Secondary Outcome: Gingival Index Level (Derived From an Average Over the 4 Implant Sites) at 1 Week
Description: as for outcome 13
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Simvastatin Group ( Treatment) | Control Group
Number analyzed (Participants) | 24 | 22
participants
  Gingival sscore of 0.50 | 1 | 1
  Gingival sscore of 1 | 2 | 1
  Gingival sscore of 1.25 | 17 | 17
  Gingival sscore of 1.50 | 4 | 3
  Gingival sscore of 1.75 | 0 | 0
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment) vs Control Group; Test type: Superiority; p = 1, Fisher Exact

16. Secondary Outcome: Probing Depth Level (Averaged Over 6 Sites) at Baseline
Description: Depth will be measured by a calibrated periodontal probe at 6 different locations, Mesiobuccal, Mid Buccal, Distobuccal, Disto Lingual, Mid Lingual and Mesio Lingual. The longitudinal course will be characterized with respect to the categorical outcome, presence of any bleeding on probing, with initial emphasis being placed upon transition approaches, with specific attention given to shifts from clinically unacceptable to clinically acceptable designations.
  probing depth is considered variable from one person to the other however a decrease or a shallower probing depth overtime is gererally seen as an improvement , thus any decrease in probing depth would be seen as signs of healing.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Simvastatin Group ( Treatment) | Control Group
Number analyzed (Participants) | 24 | 22
participants
  Probing Depth Score 1 | 0 | 1
  Probing Depth Score 2 | 3 | 5
  Probing Depth 3 | 9 | 10
  Probing Depth 4 | 9 | 6
  Probing Depth 5 | 3 | 0
  Probing Depth 6 | 0 | 0
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment) vs Control Group; Test type: Superiority; p = 0.062, Fisher Exact

17. Secondary Outcome: Probing Depth Level (Averaged Over 6 Sites) at 24 Hours
Description: as for outcome 16
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Simvastatin Group ( Treatment) | Control Group
Number analyzed (Participants) | 24 | 22
participants
  Probing Depth Score 1 | 1 | 0
  Probing Depth Score 2 | 5 | 5
  Probing Depth 3 | 7 | 10
  Probing Depth 4 | 8 | 6
  Probing Depth 5 | 2 | 1
  Probing Depth 6 | 1 | 0
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment) vs Control Group; Test type: Superiority; p = 0.54, Fisher Exact

18. Secondary Outcome: Probing Depth Level (Averaged Over 6 Sites) at 1 Week
Description: as for outcome 16
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Simvastatin Group ( Treatment) | Control Group
Number analyzed (Participants) | 24 | 22
participants
  Probing Depth Score 1 | 1 | 0
  Probing Depth Score 2 | 4 | 4
  Probing Depth 3 | 8 | 13
  Probing Depth 4 | 7 | 3
  Probing Depth 5 | 4 | 2
  Probing Depth 6 | 0 | 0
Statistical Analysis 1: Comparison: Simvastatin Group ( Treatment) vs Control Group; Test type: Superiority; p = 0.34, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Test Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03400475/Prot_000.pdf